CLINICAL TRIAL: NCT01900171
Title: A Phase I, Double-blind, Placebo-controlled, Ascending Single-dose, Safety, Tolerability and Pharmacokinetic Study of QGC001 in Healthy Male Subjects.
Brief Title: Phase I Study in Healthy Male Subjects Comparing QGC001 to Placebo
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Quantum Genomics SA (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple
Other Study IDs: QGC001/1QG1
Record Dates: First submitted 2013-06-26; First posted 2013-07-16 (Estimated); Last update posted 2013-07-16 (Estimated); Status verified 2013-07

CONDITIONS: Essential Hypertension
MeSH Terms: conditions — Essential Hypertension

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (9):
- 10 mg of QGC001 (Experimental): Each dose of QGC001 was administered orally with 100 mL of sterile water for irrigation at 08:00 in the morning of Day 1.
  Interventions: Drug: QGC001 [(3S,3'S)-4,4'-dithiobis (3-aminobutane-1-sulfonic acid)]
- 50 mg of QGC001 (Experimental): Each dose of QGC001 was administered orally with 100 mL of sterile water for irrigation at 08:00 in the morning of Day 1.
  Interventions: Drug: QGC001 [(3S,3'S)-4,4'-dithiobis (3-aminobutane-1-sulfonic acid)]
- 125 mg of QGC001 (Experimental): Each dose of QGC001 was administered orally with 100 mL of sterile water for irrigation at 08:00 in the morning of Day 1.
  Interventions: Drug: QGC001 [(3S,3'S)-4,4'-dithiobis (3-aminobutane-1-sulfonic acid)]
- 250 mg of QGC001 (Experimental): Each dose of QGC001 was administered orally with 100 mL of sterile water for irrigation at 08:00 in the morning of Day 1.
  Interventions: Drug: QGC001 [(3S,3'S)-4,4'-dithiobis (3-aminobutane-1-sulfonic acid)]
- 500 mg of QGC001 (Experimental): Each dose of QGC001 was administered orally with 100 mL of sterile water for irrigation at 08:00 in the morning of Day 1.
  Interventions: Drug: QGC001 [(3S,3'S)-4,4'-dithiobis (3-aminobutane-1-sulfonic acid)]
- 750 mg of QGC001 (Experimental): Each dose of QGC001 was administered orally with 100 mL of sterile water for irrigation at 08:00 in the morning of Day 1.
  Interventions: Drug: QGC001 [(3S,3'S)-4,4'-dithiobis (3-aminobutane-1-sulfonic acid)]
- 1,000 mg of QGC001 (Experimental): Each dose of QGC001 was administered orally with 100 mL of sterile water for irrigation at 08:00 in the morning of Day 1.
  Interventions: Drug: QGC001 [(3S,3'S)-4,4'-dithiobis (3-aminobutane-1-sulfonic acid)]
- 1,250 mg of QGC001 (Experimental): Each dose of QGC001 was administered orally with 100 mL of sterile water for irrigation at 08:00 in the morning of Day 1.
  Interventions: Drug: QGC001 [(3S,3'S)-4,4'-dithiobis (3-aminobutane-1-sulfonic acid)]
- Placebo (Placebo Comparator): The placebo was administered orally with 100 mL of sterile water for irrigation at 08:00 in the morning of Day 1.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: QGC001 [(3S,3'S)-4,4'-dithiobis (3-aminobutane-1-sulfonic acid)]
  Arms: 1,000 mg of QGC001; 1,250 mg of QGC001; 10 mg of QGC001; 125 mg of QGC001; 250 mg of QGC001; 50 mg of QGC001; 500 mg of QGC001; 750 mg of QGC001
Drug: Placebo — Contains magnesium stearate, silica dental type, anhydrous lactose
  Arms: Placebo

SUMMARY:
QGC001/1QG1 is a Phase I "first time in man" study aiming to determine the overall safety and tolerability of single ascending oral doses of QGC001 in healthy male subjects compared to placebo, as well as the pharmacokinetics of QGC001 and its metabolite EC33 and the pharmacodynamic properties of QGC001 (effects on the renin-angiotensin-aldosterone system, blood pressure and heart rate) in healthy male subjects.

ELIGIBILITY:
Inclusion Criteria:

* Caucasian, male healthy subjects of 18 to 45 years of age.
* Body weight ≥50 kg, with a body mass index calculated as weight in kg/(height in m2) from 18 to 27 kg/m2 at screening.
* Subjects will sign and date an informed consent form before any study-specific screening procedure is performed.
* Healthy, as determined by the investigator on the basis of medical history, physical examination findings, clinical laboratory test results, vital sign measurements, and digital 12 lead ECG readings.
* Non-smoker or smoker of fewer than 5 cigarettes per day as determined by history. Must be able to abstain from smoking during the inpatient stay.
* Have a high probability for compliance with and completion of the study.

Exclusion Criteria:

* Any significant cardiovascular, hepatic, renal, respiratory, gastrointestinal, endocrine, immunologic, dermatological, haematological, neurologic, psychiatric disease or history of any clinically important drug allergy.
* Acute disease state within 7 days before study day 1.
* History of drug abuse within 1 year before study day 1.
* History of alcoholism within 1 year before day 1. Consumption of more than 50 g of ethanol per day.
* Positive serologic findings for human immunodeficiency virus antibodies, hepatitis B surface antigen, and/or hepatitis C virus antibodies.
* Positive findings of urine drug screen (e.g., amphetamines, barbiturates, benzodiazepines, cannabinoids, cocaine, methadone, opiates, MDMA)
* History of any clinically important drug allergy.
* Prohibited Treatments: use of any investigational drug within 90 days or prescription drug within 30 days before investigational medical product administration.
* Consumption of any caffeine-containing products in excess of 6 cups per day (or equivalent), of grapefruit, grapefruit-containing products, or alcoholic beverages within 24 hours before study day 1.
* Use of any over-the-counter drugs including herbal supplements (except for the occasional use of acetaminophen [paracetamol], aspirin and vitamins ≤100% recommended daily allowance) within 7 days before investigational medicinal product administration.
* Donation of blood (i.e. 450 ml) within 90 days before study day 1.

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 56 (Actual)
Dates: Start 2012-02; Primary Completion 2012-05 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
Adverse events | up to 11 days
Blood pressure | up to 11 days
Heart rate | up to 11 days
Body temperature | up to 11 days
12-lead ECG | up to 11 days
Red blood cell count | up to 11 days
Haemoglobin | up to 11 days
Haematocrit | up to 11 days
White blood cell count with differential | up to 11 days
Platelet count | up to 11 days
Plasma sodium | up to 11 days
Plasma potassium | up to 11 days
Plasma calcium | up to 11 days
Plasma total bilirubin | up to 11 days
Plasma conjugated bilirubin | up to 11 days
Plasma Aspartate Amino Transferase (ASAT) | up to 11 days
Plasma Alanine Amino Transferase (ALAT) | up to 11 days
Plasma Gamma Glutamyl Transferase (GGT) | up to 11 days
Plasma alkaline phosphatases | up to 11 days
Plasma total protein | up to 11 days
Plasma Creatine PhosphoKinase (CPK) | up to 11 days
Plasma creatinine | up to 11 days
Plasma glucose | up to 11 days
Plasma cholesterol | up to 11 days
Plasma triglycerides | up to 11 days
Urinary pH | up to 11 days
Urinary protein | up to 11 days
Urinary glucose | up to 11 days
Urinary leukocytes | up to 11 days
Urinary nitrites | up to 11 days
Urinary ketones | up to 11 days
Urinary blood | up to 11 days

SECONDARY OUTCOMES:
Maximum observed plasma concentration (Cmax) of QGC001 | H0, H 0.5, H1, H1.5, H2, H3, H4, H5, H6, H9, H12, H24 and H48 post-dose
Time at which Cmax is observed (tmax) of QGC001 | H0, H 0.5, H1, H1.5, H2, H3, H4, H5, H6, H9, H12, H24 and H48 post-dose
Elimination rate constant (λz) of QGC001 | H0, H 0.5, H1, H1.5, H2, H3, H4, H5, H6, H9, H12, H24 and H48 post-dose
Terminal half-life (t1/2,z) of QGC001 | H0, H 0.5, H1, H1.5, H2, H3, H4, H5, H6, H9, H12, H24 and H48 post-dose
Area Under the Concentration-time curve (AUClast and AUC0-∞) of QGC001 | H0, H 0.5, H1, H1.5, H2, H3, H4, H5, H6, H9, H12, H24 and H48 post-dose
Maximum observed plasma concentration (MRCmax) of metabolic ratios | H0, H 0.5, H1, H1.5, H2, H3, H4, H5, H6, H9, H12, H24 and H48 post-dose
Area Under the Concentration-time curve (MRAUC) of metabolic ratios | H0, H 0.5, H1, H1.5, H2, H3, H4, H5, H6, H9, H12, H24 and H48 post-dose
Cumulative amount eliminated (Ae) | H-12 to H0 pre-dose and H0- H6, H6-H12 and H12-H24 post-dose
Fraction recovered (Fe) | H-12 to H0 pre-dose and H0- H6, H6-H12 and H12-H24 post-dose
Renal clearance (CLR) | H-12 to H0 pre-dose and H0- H6, H6-H12 and H12-H24 post-dose
Plasma renin | H-1 pre-dose and H2, H4 and H9 post-dose
  Determination of renin in blood samples. In dose groups 1 and 2, no pharmacodynamic evaluations will be done.
Plasma aldosterone | H-1 pre-dose and H2, H4 and H9 post-dose
  Determination of aldosterone in blood samples. In dose groups 1 and 2, no pharmacodynamic evaluations will be done.
Plasma cortisol | H-1 pre-dose and H2, H4 and H9 post-dose
  Determination of cortisol in blood samples. In dose groups 1 and 2, no pharmacodynamic evaluations will be done.
Plasma copeptin | H-1 pre-dose and H2, H4 and H9 post-dose
  Determination of copeptin in blood samples (if possible, will be determined later). In dose groups 1 and 2, no pharmacodynamic evaluations will be done.
Urinary aldosterone | H-12 to H0 pre-dose, H0-H6, H6-H12 and H12-H24 post-dose
  Aldosterone analysis in urine samples. In dose groups 1 and 2, no pharmacodynamic evaluations will be done.
Urinary cortisol | H-12 to H0 pre-dose, H0-H6, H6-H12 and H12-H24 post-dose
  Cortisol analysis in urine samples. In dose groups 1 and 2, no pharmacodynamic evaluations will be done.
Urinary creatinin | H-12 to H0 pre-dose, H0-H6, H6-H12 and H12-H24 post-dose
  Creatinin analysis in urine samples. In dose groups 1 and 2, no pharmacodynamic evaluations will be done.

CONTACTS AND LOCATIONS:
Locations (1):
- Biotrial PARIS, Rueil-Malmaison, France

REFERENCES:
- [Derived] Khosla J, Aronow WS, Frishman WH. Firibastat: An Oral First-in-Class Brain Aminopeptidase A Inhibitor for Systemic Hypertension. Cardiol Rev. 2022 Jan-Feb 01;30(1):50-55. doi: 10.1097/CRD.0000000000000360. PMID 33027067